CLINICAL TRIAL: NCT05568602
Title: Determination of Appropriate Limit Value for Low Dose Dexamethasone Suppression Test in Patients With Chronic Renal Failure
Brief Title: Appropriate Limit Value for 1 mg DST in Patients With Chronic Renal Failure
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: OzlemUstay3
Record Dates: First submitted 2022-10-02; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Cushing Syndrome
Keywords: cushing, dexamethasone suppression test, chronic renal failure
MeSH Terms: conditions — Cushing Syndrome; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GFR<30 ml/min: Patients screened for hypercortisolism and GFR<30ml/min
  Interventions: Diagnostic Test: Dexamethasone suppression test
- GFR>30 ml/min: Patients screened for hypercortisolism and GFR>30ml/min
  Interventions: Diagnostic Test: Dexamethasone suppression test

INTERVENTIONS:
Diagnostic Test: Dexamethasone suppression test — 1 mg Dexamethasone overnight suppression test for screening of hypercortisolism

SUMMARY:
In this study, we aimed to determine a specific cut-off value for 1mg DST to prevent false positivity usually seen in CRF patients according to the standard cut-off value of 1.8 mcg/dl.

DETAILED DESCRIPTION:
Chronic renal failure (CRF) can cause false positivity of overnight 1 mg dexamethasone suppression test (1 mg DST) in whom suspicious for Cushing Syndrome due to variability in dexamethasone bioavailability, increased cortisol secretion, disruption of diurnal rhythm, imbalance in free and bound cortisol levels because of decreased protein levels in CRF patients. In this study, we aimed to determine a specific cut-off value for 1mg DST to prevent false positivity usually seen in CRF patients according to the standard cut-off value of 1.8 mcg/dl.

The data of 1038 patients who applied to Marmara University endocrinology outpatient clinic between January 01, 2018, and December 31, 2019, and who were asked for 1 mg DST were retrospectively scanned from the hospital information and management system. The patients were divided into 4 groups according to their glomerular filtration rates (GFR). 1 mg DST results were evaluated according to GFR and ROC analysis was applied to determine the new limit value for the group whose GFR < 30 ml/min / 1.73m2 In patients classified as Group IV (the patient's GFR below 30 ml/min / 1.73m2) both 1 mg DST median and Pseudocushing Syndrome incidence were significantly higher than in other groups. The new cut-off value was found to be 3.2 mcg/dl with 100% Sensitivity and 92% specificity.

This is the first study determining a specific limit value for 1 mg DST in CRF patients with GFR below 30 ml/min / 1.73m2 to avoid false positivity in these patients. Further studies are needed in more patients on hemodialysis to check the clinically more accurate 1 mg DST cutoff value in this specific population.

ELIGIBILITY:
Inclusion Criteria:

* Between 01 January 2018 and 31 December 2019, 2173 patients who were admitted to the outpatient clinic of our hospital's Endocrine and Metabolic Diseases Department and requested 1 mg DST were included in the screening.

Exclusion Criteria:

* Being under 18 years of age
* Liver cirrhosis and /or 3-fold or more increase in liver enzymes
* Use of drugs known to interact with dexamethasone (psychotropic agents, oral contraceptives, anti-epileptic drugs, barbiturates, etc.)
* An adrenal nodule or pituitary adenoma is detected, but it is at the stage of evaluation whether it is functional or not
* Typical CS clinical findings (such as Purple stria, Buffalo Hump, moon face)
* Having an adrenal nodule or pituitary adenoma and being followed by an external center
* Lack of access to be analyzed information in the study: Albumin, AST, ALT, creatine, white blood cell (WBC), C-Reactive Protein (CRP), glycosylated hemoglobin percentage (HBA1c), glucose, sodium, potassium, thyroid stimulating hormone (TSH), body mass index (BMI), known disease and drug use information, lipid profile tests and information, lack of access to the patient's previous data
* Having a diagnosis of severe major depression
* Previously diagnosed with Cushing Syndrome or operated with this diagnosis
* Prominent hypoalbuminemia (albumin <3 g / dl)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Between 01 January 2018 and 31 December 2019, 2173 patients who were admitted to the outpatient clinic of our hospital's Endocrine and Metabolic Diseases Department and requested 1 mg DST were included in the screening.
Sampling Method: Non-Probability Sample
Enrollment: 1034 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
cut-off value for DST | 1 year
  to determine specific cut point for 1mg DST in chronic renal failure

CONTACTS AND LOCATIONS:
Overall Officials: Özlem ÜSTAY, Study Director — Marmara University
Locations (1):
- Özlem ÜSTAY, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No